CLINICAL TRIAL: NCT01236235
Title: A Non Comparative Observational Study to Describe the Duration and Outcome of Treatment in Therapy naïve HIV Positive Patients Initiated on Atazanavir (ATV)/ Ritonavir (RTV)-Based Highly Active Antiretroviral Therapy (HAART) Regimens
Brief Title: Study on Long Term Outcomes of Atazanavir in Antiretroviral-naïve Human Immunodeficiency Virus (HIV) Patients in Real Life Setting
Acronym: REMAIN
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: PharmaNet (Industry)
Responsible Party: Sponsor
Other Study IDs: AI424-401
Record Dates: First submitted 2010-11-05; First posted 2010-11-08 (Estimated); Last update posted 2013-09-05 (Estimated); Status verified 2013-09

CONDITIONS: HIV

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ARV-naïve HIV patients initiated on ATV/RTV-based therapy: Anti-retroviral (ARV)-naïve HIV patients initiated on ATV/RTV-based therapy between 2008-2010
  One cohort being observed for 3 different countries

SUMMARY:
The purpose of this study is to describe long term (> 96 weeks) efficacy and safety of Atazanavir-based regimens in real life setting.

DETAILED DESCRIPTION:
Time perspective: Collection of historical data and longitudinal follow up. Patients will be enrolled in 2011/2012 but data will be collected from medical charts from ATV initiation date (Feb 2008 - July 2010) until July 2013 at the latest (if no ATV discontinuation, or death, or lost to follow up).

Non probability sample:

* Specialized HIV management centers will be contacted in order to recruit about 15-20 sites per country.
* Each site will have to enroll an average of 8-12 consecutive patients (min:5; max:30) fulfilling the inclusion/exclusion criteria.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female HIV patients ≥ 18 years old at ATV/RTV initiation treatment date
* Outpatient seen in routine consultation whatever the reason, between January 1st 2011 and March 31st 2012
* Commencing an ATV/RTV-based regimen including at least 2 nucleoside reverse transcriptase inhibitors (NRTI) after February 1st 2008 and before July 31st 2010, regardless of the current ARV treatment ongoing at enrollment visit

Exclusion Criteria:

* Patient exposed to or who began ATV/RTV prior to February 1st 2008, or after July 31st 2010 or without a known start date for ATV/RTV therapy
* Exposure to more than 4 weeks of any ARV prior to initiation of ATV/RTV treatment
* Participation in a clinical trial with ATV at the time of or after initiation of ATV/RTV-based regimen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients attending HIV specialized management centers will be considered.
Sampling Method: Non-Probability Sample
Enrollment: 525 (Actual)
Dates: Start 2011-01; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Proportion of patients remaining on ATV-based treatment over time | Up to 5.5 years
  Every 6 months from ATV initiation till July 2013 at the latest (maximum follow-up time up to 5.5 years)

SECONDARY OUTCOMES:
Time to discontinuation of ATV | Every 6 months up to 5.5 years
Reasons for ATV discontinuation | Every 6 months up to 5.5 years
Percent of patients with HIV-1 ribonucleic acid (RNA) < 50 and < 500 c/mL | Every 6 months up to 5.5 years
Mean change in HIV-1 RNA | Every 6 months up to 5.5 years
Time to viral failure (HIV-1 RNA ≥ 50 and ≥ 500 c/mL) | Every 6 months up to 5.5 years
Mean change in Cluster of differentiation 4 (CD4) cell count | Every 6 months up to 5.5 years
Adverse events (AEs) related to ATV | Every 6 months up to 5.5 years
Lipid profile | Every 6 months up to 5.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (38):
- Germany (10):
  - Local Institution, Aachen
  - Local Institution, Berlin
  - Local Institution, Düsseldorf
  - Local Institution, Freiburg im Breisgau
  - Local Institution, Hamburg
  - Local Institution, Hanover
  - Local Institution, Mannheim
  - Local Institution, München
  - Local Institution, Regensburg
  - Local Institution, Stuttgart
- Portugal (9):
  - Local Institution, Aveiro
  - Local Institution, Barreiro
  - Local Institution, Lisbon
  - Local Institution, Portimão
  - Local Institution, Porto
  - Local Institution, Pragal
  - Local Institution, Santarém
  - Local Institution, São Martinho do Bispo
  - Local Institution, Vila Nova de Gaia
- Spain (19):
  - Local Institution, Alcorcón
  - Local Institution, Badalona
  - Local Institution, Barcelona
  - Local Institution, Granada
  - Local Institution, Granollers
  - Local Institution, Guadalajara
  - Local Institution, Jerez de la Frontera
  - Local Institution, Leganés
  - Local Institution, Logroño
  - Local Institution, Madrid
  - Local Institution, Marbella
  - Local Institution, Mataró
  - Local Institution, Málaga
  - Local Institution, Móstoles
  - Local Institution, Santiago de Compostela
  - Local Institution, Seville
  - Local Institution, Tarragona
  - Local Institution, Valencia
  - Local Institution, Zaragoza

REFERENCES:
- [Derived] Teofilo E, Rocha-Pereira N, Kuhlmann B, Antela A, Knechten H, Santos J, Jimenez-Exposito MJ; REMAIN study group. Long-Term Efficacy, Tolerability, and Renal Safety of Atazanavir/Ritonavir-based Antiretroviral Therapy in a Cohort of Treatment-Naive Patients with HIV-1 Infection: the REMAIN Study. HIV Clin Trials. 2016 Feb;17(1):17-28. doi: 10.1080/15284336.2015.1112494. PMID 26899539
- See also: BMS Clinical Trials Disclosure — http://www.bms.com/clinical_trials/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx
- See also: For FDA Safety Alerts and Recalls refer to the following link: http://www.fda.gov/MEDWATCH/safety.htm — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm